CLINICAL TRIAL: NCT03839784
Title: Building a Platform for Precision Anesthesia in the Geriatric Surgical Patient
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David R. Drover, Professor of Anesthesiology, Stanford University
Other Study IDs: 55169
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Decline; Cognitive Change; Cognitive Impairment; Postoperative Delirium; Anesthesia; Reaction; Anesthesia; Adverse Effect
MeSH Terms: conditions — Cognitive Dysfunction; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neurocognitive Assessment Arm
  Interventions: Combination Product: Neurocognition Interventions

INTERVENTIONS:
Combination Product: Neurocognition Interventions — EEG, Neurocognitive Battery Testing, and Immune Profiles

SUMMARY:
The research team is creating a foundational infrastructure in order to develop a precision medicine approach for geriatric patients who require surgery with anesthesia. The team plans to build the first of its kind comprehensive database of demographic and risk factor questionnaire responses, biobanked blood specimens, intraoperative electroencephalography (EEG), and inclusive cognitive testing throughout patient interaction starting at the preop appointment until a year later. This will be used to create a predictive model of periooperative neurocognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old (inclusive)
* Non cardiac general elective surgery
* General anesthesia is expected for 2+ hours

Exclusion Criteria:

* Alzheimer's
* Dementia
* Parkinson's
* History of neurodegenerative diseases
* Medication for depression (ie. Benzodiazepines)
* Alcoholism
* Discretion of PI

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Stanford Hospital geriatric patients having surgery.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Neurocognitive Disorders | 3 years
  Neurocognitive Assessment Battery

CONTACTS AND LOCATIONS:
Overall Officials: David Drover, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided